CLINICAL TRIAL: NCT06532305
Title: The Effects of Empowerment Classes on Burnout Syndrome and Emotional Stress Among Southeast Asian Migrant Care Workers: A Randomized Crossover Study
Brief Title: Helping Overcome Pressure and Exhaustion: Empowerment Classes for Southeast Asian Migrant Care Workers
Acronym: HOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 202406135RINE
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Heart Rate Variability; Burnout; Depression
Keywords: empowerment; burnout; dementia; migrant care worker
MeSH Terms: conditions — Burnout, Psychological; Depression; Empowerment; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowerment classes (Experimental): Content:
  Mental Health and Stress Management: Techniques and strategies for managing stress, mindfulness practices, and mental health awareness.
  Dementia Care Skills: Training on dementia care, communication with dementia patients, and specific caregiving techniques.
  Language and Communication Skills: Improving proficiency in local languages and enhancing communication skills relevant to caregiving.
  Follow-up: After completing the empowerment classes, participants will switch to the social gatherings intervention.
  Interventions: Behavioral: HOPE empowerment classes
- Social gatherings (Active Comparator): Content:
  Social Interaction: Regular gatherings to promote social bonding and peer support among care workers.
  Recreational Activities: Group activities designed to foster relaxation and social engagement.
  Informal Discussions: Opportunities for care workers to share experiences and coping strategies in an informal setting.
  Follow-up: After completing the social gatherings, participants will switch to the empowerment classes intervention.
  Interventions: Behavioral: HOPE empowerment classes

INTERVENTIONS:
Behavioral: HOPE empowerment classes — A three-month empowerment course.

SUMMARY:
As Taiwan's population ages, Southeast Asian migrant care workers are widely employed to fill the care labor gap. These workers often face symptoms of burnout and emotional stress due to long working hours and high-pressure environments. This study aims to evaluate the effects of empowerment classes on reducing burnout symptoms and emotional stress among Southeast Asian migrant care workers. The empowerment classes are designed based on expert consensus and cover three core areas: mental health and stress management, dementia care skills, and language and communication skills. The curriculum is tailored to the practical needs and cultural backgrounds of the migrant workers. A total of 120 Indonesian care workers will be randomly assigned to two groups. The first group will undergo a three-month empowerment course, while the second group will initially participate in social gatherings. Afterward, the groups will switch interventions. The study will last for 12 months, and each participant will complete seven assessments, including heart rate variability measurements and online questionnaires. The questionnaires will include the Patient Health Questionnaire-2 (PHQ-2), the Copenhagen Burnout Inventory (CBI), the Life and Cultural Adaptation Questionnaire, and the Language Proficiency Questionnaire. The study anticipates that the empowerment classes will reduce burnout symptoms and emotional stress, while enhancing cultural adaptation and language proficiency among migrant care workers.

DETAILED DESCRIPTION:
Study Design:

The study employs a randomized crossover design involving 120 Indonesian care workers in Taiwan. Participants will be randomly assigned to two groups. The first group will undergo a three-month empowerment course initially, while the second group will participate in social gatherings. After three months, the interventions will be switched between the groups. The empowerment classes will cover three core areas: mental health and stress management, dementia care skills, and language and communication skills, tailored to the workers' practical needs and cultural backgrounds.

Duration:

The study will last for 12 months, starting from July 26, 2024, to July 25, 2025.

Data Collection:

Participants will complete seven assessments, including heart rate variability measurements and online questionnaires. The questionnaires will include the Patient Health Questionnaire-2 (PHQ-2), the Copenhagen Burnout Inventory (CBI), the Life and Cultural Adaptation Questionnaire, and the Language Proficiency Questionnaire.

Expected Outcomes:

The study anticipates that the empowerment classes will reduce burnout symptoms and emotional stress, while enhancing cultural adaptation and language proficiency among migrant care workers.

Ethical Considerations:

Participation in this study is voluntary, and participants can withdraw at any time without negative consequences. All personal data will be kept confidential and used solely for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Indonesian migrant care workers responsible for caring for patients in homes or care institutions.
* Aged 18 years or older.

Exclusion Criteria:

* Individuals unable to read the informed consent form or questionnaires in Indonesian.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-26 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Burnout levels | 12 months
  Measured using the Copenhagen Burnout Inventory (CBI). The primary outcome will be the change in burnout levels from baseline to the end of each intervention period. Burnout will be assessed in three domains: personal burnout, work-related burnout, and client-related burnout. Higher scores on the CBI indicate a higher level of burnout, meaning worse outcomes in terms of burnout severity. The range of CBI is 0-100.
Emotional Stress | 12 months
  Measured using the Patient Health Questionnaire-2 (PHQ-2). The outcome will be the change in emotional stress levels from baseline to the end of each intervention period. A PHQ-2 score ranges from 0-6. Higher scores on the PHQ-2 indicate greater severity of depressive symptoms, meaning worse outcomes in terms of emotional stress.
Heart Rate Variability | 12 months
  Heart Rate Variability measurements will be used to assess changes in autonomic nervous system function, providing an objective measure of stress levels.

SECONDARY OUTCOMES:
Cultural Adaptation | 12 months
  Measured using the Life and Cultural Adaptation Questionnaire. The secondary outcome will be the change in cultural adaptation levels from baseline to the end of each intervention period. There is a total of 11 questions that inquire about the respondent's adaptation to daily life, work, and culture in Taiwan. Its total score ranges from 11-66. Each item is rated on a scale of 1 to 6, with higher scores indicating better adaptation.
Language Proficiency | 12 months
  Assessed using the Language Proficiency Questionnaire. The secondary outcome will be the change in language proficiency levels from baseline to the end of each intervention period. There is a total of 7 questions primarily aimed at understanding the current usage of Mandarin and Taiwanese. Each item is rated on a scale of 1 to 6, with higher scores indicating better communication skills in the respective language. The total score ranges from 7 to 42.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No